CLINICAL TRIAL: NCT04741646
Title: Phosphate Binder Therapy and Chronic Kidney Disease in Children
Brief Title: Ferric Citrate and Chronic Kidney Disease in Children
Acronym: FIT4KID
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: University of California, Los Angeles (Other)
Collaborators: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Principal Investigator, Isidro Salusky, MD, Distinguished Professor of Pediatrics at the David Geffen School of Medicine at UCLA, Chief of Pediatric Nephrology and Director of the Pediatric Dialysis Program, University of California, Los Angeles
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: U01DK122013 (NIH); 1U01DK122013 (NIH); 22-001133 (Other: UCLA IRB)
Record Dates: First submitted 2021-02-02; First posted 2021-02-05 (Actual); Last update posted 2025-05-02 (Actual); Status verified 2025-04

CONDITIONS: Chronic Kidney Diseases
Keywords: Pediatric; CKD; Phosphate Binder
MeSH Terms: conditions — Renal Insufficiency, Chronic | interventions — ferric citrate

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Treatment Arm (Experimental): During the 12-month trial, participants will be given a fixed weight-based dose of Ferric Citrate (FC). The full medication dose will be 3g/day for participants weighing <31 kg, 5g/day for those weighing >31 - <51 kg, and 6g/day for participants >51 kg. These doses will be divided into three doses to be taken with meals.
  Interventions: Drug: Ferric Citrate
- Control Arm (Placebo Comparator): During the 12-month trial, participants will be given a fixed weight-based dose of Placebo. The full medication dose will be 3g/day for participants weighing <31 kg, 5g/day for those weighing >31 - <51 kg, and 6g/day for participants >51 kg. These doses will be divided into three doses to be taken with meals.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Ferric Citrate — Auryxia® 210 mg ferric iron tablets equivalent to 1 g of FC will be supplied as 200 tablets in 400cc high-density polyethylene bottles.
  Other Names: Auryxia
  Arms: Treatment Arm
Drug: Placebo — Placebo to match Ferric Citrate tablets
  Arms: Control Arm

SUMMARY:
We will conduct a 12-month, double-blind, randomized, placebo-controlled trial to assess the effects of therapy with ferric citrate (FC) on changes in intact FGF23 levels (iFGF23, primary endpoint) in 160 pediatric patients (80 in each of the two arms) aged 6-18 years of either sex with chronic kidney disease (CKD) stages 3-4 and age-appropriate normal serum phosphate levels. Participants will be randomized to one of the two groups: 1) FC or 2) FC placebo. Participants will be recruited from 20 core clinical sites.

DETAILED DESCRIPTION:
We will conduct a double-blind, randomized, placebo-controlled trial to assess the effects of therapy with ferric citrate (FC) on changes in intact FGF23 levels (iFGF23, primary endpoint) aged 6-18 years of either sex with chronic kidney disease (CKD) stages 3-4 and age-appropriate normal serum phosphate levels. Participants will be randomized to one of the two groups: 1) FC or 2) FC placebo. Participants will be recruited from 20 core clinical sites.

Schedule of Intervention: During the 12-month trial, participants will be given a daily fixed weight-based dose of FC.

Schedule for data collection/analyses to be performed:

Blood for primary outcome assessments will be collected at screening, baseline and at months 3, 6, 9, 12. Blood for safety assessments will be collected at the the months 1, 2, 3, 6, 9, 12.

The primary analyses for this 2-arm trial will compare log-transformed iFGF23 values over 12 months between the treatment and the placebo arms. The analysis will use a linear mixed-effects model, including stratification factors CKD stage and urine protein to creatinine ratio, with random participant effects accounting for repeated measurements, and a fixed treatment effect, which interacts with a time indicator (Months 3-12 vs. Baseline/Screening).

Primary objectives:

* To assess the effects of therapy with FC on iFGF23 levels
* To determine safety and tolerability of FC.

Secondary objectives:

• To assess the effects of FC on anemia and indices of mineral and bone metabolism.

Primary Endpoint:

• iFGF23 level

Safety and Tolerability Endpoints:

• Ability to safely tolerate FC

Secondary Endpoints:

* Anemia
* Indices of mineral and bone metabolism

This is a Phase 2 study with participation from 20 sites that will take 36 months to complete enrollment and a total of 48 months to complete data collection with each participant being part of the study for 12 months.

Study website: fit4kid.dgsom.ucla.edu

ELIGIBILITY:
Inclusion Criteria:

1. Ages 6 to 18 years (inclusive);
2. Estimated Glomerular Filtration Rate (GFR) of 15-59 ml/min per 1.73 m2 by modified Chronic Kidney disease in Children (CKiD) under 25 (U25) formula;56
3. Serum phosphate <=5.9 mg/dl;
4. Serum ferritin <500 ng/ml and TSAT <50%;
5. For those patients treated with growth hormone, calcitriol, nutritional vitamin D, iron, and/or erythropoiesis-stimulating agents (ESAs) such treatments must have stable dosing for at least 2 weeks prior to screening;
6. Able to swallow tablets;
7. Able to eat at least two meals a day;
8. In the opinion of the investigator, willing and able to follow the study treatment regimen and comply with the site investigator's recommendations.

Exclusion Criteria:

1. Patients currently treated with phosphate binders.
2. History of allergy to all ingredients (including non-medical ingredients) in both products (i.e. investigational product and placebo)
3. Current intestinal malabsorption, documented in the medical record; disease, inflammatory bowel syndrome, and/or Crohn's Disease.
4. Anticipated initiation of dialysis or kidney transplantation within 6 months
5. Current or planned future systemic immunosuppressive therapy
6. Prior solid organ transplantation
7. Receipt of bone marrow transplant within two years of screening
8. Current pregnancy, lactation or female subjects who have reached menarche, unless using highly-effective contraception as outlined in section 7.1.1 of Protocol
9. Patients participating in other interventional study (observational study participation permitted)
10. Poor adherence to medical treatments in the opinion of the investigator
11. Cystinosis
12. Fanconi syndrome
13. Hemochromatosis or laboratory tests indicating possible hemochromatosis or other iron overload (primary or secondary) syndrome

Ages: 6 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 160 (Estimated)
Dates: Start 2022-06-17 (Actual); Primary Completion 2027-10 (Estimated); Study Completion 2027-10 (Estimated)

PRIMARY OUTCOMES:
iFGF23 levels | 12 months
  Compared to placebo, active treatment with FC will lower iFGF23 levels
Safety of Ferric Citrate | 12 months
  Comparing proportion of subjects with AE and SAE between arms
Tolerability of Ferric Citrate | 12 months
  Compared with placebo, active treatment will be tolerable

SECONDARY OUTCOMES:
Effects on Transferrin Saturation (TSAT) | 12 months
  Compared with placebo, active treatment with FC will be associated with larger increase in hemoglobin, higher TSAT and higher Ferritin from baseline
Effects on PTH and 1,25 D | 12 months
  Compared to placebo, active treatment with FC will be associated with a larger decrease in PTH and larger increase in 1,25 D from baseline

OTHER OUTCOMES:
GFR | 12 months
  Compared to placebo, active treatment with FC will be associated with smaller decrease in GFR over time
Osteoid thickness | 12 months
  Compared to placebo, active treatment with FC will be associated with a larger decrease of osteoid thickness from baseline
Effects on bone expression | 12 months
  Compared to placebo, active treatment with FC will be associated with a greater reduction in bone expression of FGF23
Effects on phosphate | 12 months
  Compared to placebo, active treatment with FC will be associated with a greater reduction in 24 hours urinary phosphate and fractional excertion of phosphate
Effects on calcium | 12 months
  Compared to placebo, active treatment with FC will be associated with a greater incresae in serum calcium levels from baseline
Effects on 1,25 (OH) D levels | 12 months
  Compared to placebo, active treatment with FC will be associated with a greater increase from baseline in serum 1,25 (OH) D levels
Effects on bone biomarkers | 12 months
  Compared to placebo, active treatment with FC will be associated with greater reduction from baseline of bone biomarkers of turnover
Effects on Klotho | 12 months
  Compared to placebo, active treatment with FC will be associated with greater increase from baseline in levels of Klotho
Effects on cFGF23 | 12 months
  Compared to placebo, active treatment with FC will be associated with greater reduction from baseline in cFGF23

CONTACTS AND LOCATIONS:
Overall Officials: Isidro B Salusky, MD, Principal Investigator — University of California, Los Angeles
Locations (20):
- United States (18):
  - University of California, Los Angeles, Los Angeles, California
  - Children's Hospital of Orange County, Orange, California
  - University of California, San Francisco, San Francisco, California
  - Arnold Palmer Hospital for Children, Orlando, Florida
  - Emory University, Atlanta, Georgia
  - Indiana U, Indianapolis, Indiana
  - Children's Mercy Hospital, Kansas City, Kansas City, Missouri
  - Washington U, St Louis, Missouri
  - Cohen's Childrens, New York, New York
  - Children's Hospital at Montefiore, The Bronx, New York
  - Duke, Durham, North Carolina
  - Cincinnati Children's Hospital Medical Center, Cincinnati, Ohio
  - Nationwide Children's, Columbus, Ohio
  - OHSU, Portland, Oregon
  - Children's Hospital of Philadelphia, Philadelphia, Pennsylvania
  - Children's Medical Center, Dallas, Dallas, Texas
  - Baylor College of Medicine, Houston, Texas
  - UTH, Houston, Texas
- Canada (2):
  - BC Children's Hospital Research Institute, Vancouver, British Columbia
  - SickKids, Toronto, Ontario

IPD SHARING:
Plan to Share IPD: Yes
All de-identified clinical data, including study outcomes and participant characteristics will be submitted to the National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) Central Repository at the completion of the study. De-identified research samples blood and urine will also be provided to the NIDDK central reporsitory
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: the IPD will become available 12 months after study completion.
Access Criteria: Access will be provided by National Institute of Health and any researcher will be able to request access from NIH once the data becomes available.

REFERENCES:
- [Derived] Hanudel MR, Laster ML, Portale AA, Dokras A, Quigley RP, Guzman GAL, Zaritsky JJ, Hayde NA, Kaskel FJ, Mitsnefes MM, Ramirez JA, Imani PD, Srivaths PR, Kogon AJ, Denburg MR, Blydt-Hansen TD, Reyes LZ, Greenbaum LA, Weidemann DK, Warady BA, Elashoff DA, Mendley SR, Isakova T, Salusky IB. A review of ferric citrate clinical studies, and the rationale and design of the Ferric Citrate and Chronic Kidney Disease in Children (FIT4KiD) trial. Pediatr Nephrol. 2022 Nov;37(11):2547-2557. doi: 10.1007/s00467-022-05492-7. Epub 2022 Mar 2. PMID 35237863